CLINICAL TRIAL: NCT03729908
Title: Effects of an Animal Assisted Mindfulness Intervention for Patients With Acquired Brain Injury: A Randomized Controlled Trial
Brief Title: Animal Assisted Mindfulness Intervention (AAMI) for Patients With Acquired Brain Injury
Acronym: AAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Rehab Basel (Other); University of Basel (Other); University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-00564
Record Dates: First submitted 2018-09-26; First posted 2018-11-05 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-01

CONDITIONS: Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal assisted mindfulness based intervention (Experimental): The intervention is the AAMI. Trained animals that live in the "Therapie-Tiergarten" of REHAB Basel will function as therapy animals. Trained psychologists will lead the AAMI.
  Interventions: Behavioral: Animal assisted mindfulness based intervention
- Anti-stress program (Active Comparator): The active control intervention consists of the same program, however without the inclusion of animals (Anti-Stress program, ASP).
  Interventions: Behavioral: Anti-stress program

INTERVENTIONS:
Behavioral: Animal assisted mindfulness based intervention — A mindfulness based intervention in the presence of an animal
  Arms: Animal assisted mindfulness based intervention
Behavioral: Anti-stress program — A mindfulness based intervention with no reference to animals
  Arms: Anti-stress program

SUMMARY:
The aim of this study is to investigate the effect of an animal assisted mindfulness intervention (AAMI) on patients with acquired brain injuries on their global severity of psychological distress.

In addition, the effects on the patients' symptoms of depression, anxiety, perceived stress, mood, coping and mindfulness/self-compassion will be assessed.

The study experimental condition consists of 6 weeks of intervention, containing 6 different modules. In every session, an animal will be present.

In the control condition, the same program and same exercises will be used without the presence of or reference to animals. Sessions take place two times a week for 6 weeks (leading up to a total of 12 experimental/control sessions), each lasting for about 60 minutes.

24 participants are planned to be included, 12 patients in each group.

DETAILED DESCRIPTION:
It was estimated that a total sample of 24 participants (12 patients in each group) would provide enough power to detect a medium effect. Since we had several dropouts, two additional groups (one intervention and one control) were started. This lead to the inclusion of 31 participants with a total sample size of 25 participants finishing the program.

ELIGIBILITY:
Inclusion Criteria:

* Patients of REHAB Basel
* Acquired Brain Injury (ABI); FIM (Functional Independence Measure) cut-off score defined as > 60
* Depressive or/and anxiety symptoms
* Psychological difficulties coping with the actual life situation
* 18 years or older
* Willing to work with therapy animals
* German speaking
* Willingness to participate/informed consent

Exclusion Criteria:

* Communication and articulation is not possible
* Allergy to animals
* Aversion against animals
* Schizophrenic-related comorbidity
* Mobilization to "Therapietiergarten" not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
General psychological distress | 11 weeks
  Measured via BSI (Global Severity Index GSI). The Global Severity Index (GSI) is designed to help quantify a patient's severity-of-illness and provides a single composite score for measuring the outcome of a treatment program based on reducing symptom severity. Minimal total score = 0, maximal total score = 212 (higher values represent a worse outcome)

SECONDARY OUTCOMES:
Depression | 11 weeks
  Measured via BDI-FS (Beck Depression Inventory - Fast Screen for Medical Clients, without somatic items). The BDI-FS is a fast screen assessment of depression for medical patients. The minimum score is 0, the maximum score is 21, higher values represent a worse outcome.
Perceived Stress | 11 weeks
  Measured via the PSS-10-D (Perceived Stress Scale - 10). The Perceived Stress Scale was developed to measure the degree to which situations in one's life are appraised as stressful. The minimal total score is 1, the maximal total score is 40. Higher values represent worse outcome.
Mindfulness | 11 weeks
  Measured via the FFA-14 (Freiburger Fragebogen zur Achtsamkeit). Minimum total score is 0, maximum total score is 39. Higher values represent a better outcome.
Self-compassion | 11 weeks
  Measured via SCS-D Kurzversion (Self-compassion scale - Deutsch): Minimum total score is 1, maximum total score is 60, higher values represent a better outcome.
Coping | 11 weeks
  Measured via Brief COPE-G: The Brief COPE (-G, German version) Inventory is a multidimensional coping inventory to assess the different ways in which people respond to stress. It measures problem-focused coping, emotion-focused coping, and dysfunctional coping. Each subscale ranges between 1 and 8 with higher values representing higher scores in the respective coping strategy.
Visual Analogue Scale (VAS) | 11 weeks
  A VAS measuring motivation, emotion, cognition and attitude towards animals. The Visual Analogue Scales (VAS) provide a simple technique for measuring subjective experience and are continuous scales comprised of a horizontal line. Minimum score for each item is 0, maximum score is 160 with higher scores representing better outcomes.
Mood | 6 weeks
  Measured via the MDBF before and after each session: Mehrdimensionaler Befindlichkeitsfragebogen. The "Mehrdimensionaler Befindlichkeitsfragebogen" (MDBF) is a German-language instrument to assess the 3 mood dimensions pleasant-unpleasant, awake-sleepy, calm-restless and includes 24 items. Minimum score is 4, maximum score is 20.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Hediger, Principal Investigator — University of Basel
Locations (1):
- REHAB Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided